CLINICAL TRIAL: NCT06986200
Title: MultiCPR: The Influence of Firefighter's PPE on Chest Compressions
Brief Title: MultiCPR: The Influence of Firefighter's PPE on Chest Compressions (MultiCPR3)
Acronym: MultiCPR3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Mathias Maleczek, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: MultiCPR_3
Record Dates: First submitted 2025-05-13; First posted 2025-05-22 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Cardiac Arrest (CA); Occupational Health
MeSH Terms: conditions — Heart Arrest | interventions — Chest Wall Oscillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One minute rotation intervals (Active Comparator): Chest compressions will be done with one minute rotation intervals
  Interventions: Procedure: Chest Compressions; Procedure: One minute rotation intervall
- Two minute rotation intervals (Active Comparator): Chest compressions will be done with two minute rotation intervals
  Interventions: Procedure: Chest Compressions; Procedure: Two minute rotation intervall

INTERVENTIONS:
Procedure: Chest Compressions — Performing chest compressions in full firefighter's personal protcetion equipment
Procedure: One minute rotation intervall — Chest compressions using a one minute rotation intervall
  Arms: One minute rotation intervals
Procedure: Two minute rotation intervall — Chest compressions using a two minute rotation intervall
  Arms: Two minute rotation intervals

SUMMARY:
The aim of this clinical study is to evaluate the impact of wearing firefighters' personal protective equipment (PPE) on the quality of chest compressions during simulated resuscitation scenarios. The study compares the effects of one-minute versus two-minute intervals for switching the individual performing compressions.

How does the clinical trial work? This randomized cross over trial will be conducted in several locations and will involve a total of 38 fire-fighters. The study will be conducted by the Department of Anesthesiology of the Medical University of Vienna.

Participation in this clinical study is expected to last 30 minutes in total. Participants are randomized to either one or two minute intervalls of performing chest compressions in teams of two. After a cooling-of phase of at least 24 hours, they will be switched to the other group.

Chest compressions will be performed for 12 minutes in full firefighter's PPE. Primary outcome will be chest compression depth.

ELIGIBILITY:
Inclusion:

* Healthy fire-fighters trained in CPR
* CPR Training in the last four years
* Fit and rested

Exclusion:

- Pregnant participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2025-06-16 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Chest Compressions depth | during 12 minutes of chest compressions. 2x12 = 24minutes in total per participant
  depth in milimeter

SECONDARY OUTCOMES:
Chest compression rate | during 12 minutes of chest compressions. 2x12 = 24minutes in total per participant
Incomplete recoil (leaning) during chest compressions | during 12 minutes of chest compressions. 2x12 = 24minutes in total per participant
  Incomplete recoil is an important measure during chest compressions as it impairs ventricular filling. Incomplete recoil is measured in milimeters.

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Simulation Center, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No